CLINICAL TRIAL: NCT01711541
Title: Carboplatin-Paclitaxel Induction Chemotherapy and ABT-888 (Veliparib) - a Phase 1/Randomized Phase 2 Study in Patients With Locoregionally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Combination Chemotherapy With or Without Veliparib in Treating Patients With Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02009; NCI-2012-02009 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A091101; A091101 (Other: Alliance for Clinical Trials in Oncology); A091101 (Other: CTEP); N01CM62201 (NIH); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Stage IVA Oropharyngeal Carcinoma AJCC v7; Stage IVB Oropharyngeal Carcinoma AJCC v7
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Fluorouracil; dehydroftorafur; Hydroxyurea; Paclitaxel; Taxes; Radiotherapy; Radiation; veliparib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (veliparib, combination chemotherapy) (Experimental): Patients receive veliparib PO BID on days 1-7, paclitaxel IV over 60 minutes on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients then continue on to concomitant chemoradiotherapy.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Fluorouracil; Drug: Hydroxyurea; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Radiation: Radiation Therapy; Drug: Veliparib
- Arm II (placebo, combination chemotherapy) (Experimental): Patients receive placebo PO BID on days 1-7. Patients also receive paclitaxel and carboplatin as in Phase I. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Within 10 days from completion of course 2, patients begin concomitant chemoradiotherapy.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Fluorouracil; Drug: Hydroxyurea; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Placebo Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Hydroxyurea — Given PO
  Other Names: Droxia; Hydrea; Hydroxycarbamide; Litalir; Onco-Carbide; Oncocarbide; Oxeron; SQ 1089; SQ-1089; Syrea; WR 83799
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo, combination chemotherapy)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Name of Radiation Therapy Course; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888
  Arms: Arm I (veliparib, combination chemotherapy)

SUMMARY:
This partially randomized phase I/II trial studies the side effects and best dose of veliparib when given together with combination chemotherapy and to see how well they work in treating patients with stage IV head and neck cancer. Drugs used in chemotherapy, such as docetaxel, cisplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether combination chemotherapy is more effective when given with or without veliparib in treating head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD), recommended phase II dose, dose limiting toxicity (DLT), and safety of ABT-888 (veliparib) with carboplatin and paclitaxel induction chemotherapy in locoregionally advanced head and neck (LAHNC) patients. (Phase I) II. Compare magnitude of tumor shrinkage (response) following 2 cycles of induction chemotherapy with and without ABT-888 in LAHNC. (Phase II)

SECONDARY OBJECTIVES:

I. Compare progression-free (PFS), disease-specific (DSS), and overall survival (OS) in subjects treated with or without ABT-888. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of veliparib followed by a phase II study.

PHASE I: Patients receive veliparib orally (PO) twice daily (BID) on days 1-7, paclitaxel intravenously (IV) over 60 minutes on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients then continue on to concomitant chemoradiotherapy.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive veliparib, paclitaxel, and carboplatin as in Phase I. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Within 10 days from completion of course 2, patients begin concomitant chemoradiotherapy.

ARM II: Patients receive placebo PO BID on days 1-7. Patients also receive paclitaxel and carboplatin as in Phase I. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Within 10 days from completion of course 2, patients begin concomitant chemoradiotherapy.

CONCOMITANT CHEMORADIOTHERAPY: Patients are assigned to 1 of 2 regimens of concomitant chemoradiotherapy based on the guidelines of the institution where they are being treated.

OPTION I (CONCOMITANT CHEMORADIATION WITH CISPLATIN): Patients receive cisplatin IV on days 1 and 22 and undergo radiation therapy 5 days per week for 6 weeks. Treatment repeats every 2 weeks for 5 courses.

OPTION II (CONCOMITANT CHEMORADIATION WITH TFHX): Patients receive hydroxyurea PO every 12 hours on days 1-5 for up to 11 doses, fluorouracil IV over 120 hours on days 1-5, paclitaxel IV on day 1, and undergo radiation therapy BID on days 1-5. Treatment repeats every 2 weeks for 5 courses.

After completion of study treatment, patients are followed up at 2 weeks, 1, 3, 6, 12, 18, 24, 30, 36, 48, and 60 months. Patients who progress will be followed up every 6 months through year 5.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I:
* Patients who are treatment naïve, high risk, stage IVa/IVb (all other sites) and histologically proven squamous cell carcinoma of the head and neck (SCCHN) with no definitive evidence of metastatic disease, excluding patients with oropharynx human papillomavirus (HPV)-positive tumors; in summary, those patients eligible are newly diagnosed and treatment naive:

  * Stage IVa-b squamous cell carcinoma other than oropharyngeal cancer (OPC), or
  * Oropharyngeal cancer (OPC) HPV-negative, stage IVa-b
* PHASE II:
* Patients who are treatment naïve, high risk, stage IVa/IVb (all other sites) histologically proven SCCHN with no definitive evidence of metastatic disease; in summary, those patients eligible are:

  * Stage IVa-b SCCHN other than OPC, or
  * OPC, HPV-negative, IVa-b, or
  * OPC, HPV positive, with greater than 10 pack-year smoking history and N2b-N3 disease
* PHASE I AND II:
* Patients must have at least one measurable site of disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria; i.e., patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan magnetic resonance imaging (MRI), or calipers by clinical exam
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must be able to swallow the drug
* Ability to understand and the willingness to sign a written informed consent document
* Leukocytes >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x institutional ULN as calculated by Cockcroft-Gault
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above ULN as calculated by Cockcroft-Gault
* Patients who are receiving any other investigational agents are not eligible
* Patients with active seizure or a history of seizure are not eligible
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ABT-888 or other agents used in study, including Cremophor, carboplatin, paclitaxel, cisplatin, 5-fluorouracil, hydroxyurea, or any compounds of similar chemical or biologic composition are not eligible
* Patients with impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of ABT-888 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection) are not eligible to participate in this study
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements are not eligible to participate in the study
* Pregnant women are not eligible to participate in this study; NOTE: women of child bearing potential must have a negative serum or urine pregnancy test within 7 days prior to treatment

  * Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately;
  * Breastfeeding should be discontinued if the mother is treated with ABT-888
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are not eligible
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent are not eligible to participate in this study; topical or inhaled corticosteroids are allowed
* Patients with other malignancies within the past 2 years, except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin or surgically treated early stage solid tumors are ineligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10-22 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonas De Souza, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study originally opened at Dose Level 0 with a treatment of Docetaxel, cisplatin and flouricil (TPF) in combination with ABT-888 (veliparib). With a concern for the feasibility of this regimen in other reported studies, this study was suspended and re-opened with a treatment of Carboplatin and Paclitaxel in combination with ABT-888.
Groups:
- Dose Level 0: ABT-888 doses will be given at 200 mg bid for 7 days in combination with TPF Induction
- Dose Level 0B: ABT-888 doses will be given at 200 mg bid for 7 days in combination with paclitaxel 100 mg/m2 and carboplatin AUC 6.
- Dose Level 1: ABT-888 doses will be given at 250 mg bid for 7 days in combination with paclitaxel 100 mg/m2 and carboplatin AUC 6.
- Dose Level 2: ABT-888 doses will be given at 300 mg bid for 7 days in combination with paclitaxel 100 mg/m2 and carboplatin AUC 6.
- Dose Level 3: ABT-888 doses will be given at 350 mg bid for 7 days in combination with paclitaxel 100 mg/m2 and carboplatin AUC 6.
Period: Overall Study
Arm/Group | Dose Level 0 | Dose Level 0B | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 4 | 4 | 3 | 6 | 7
Completed | 4 | 3 | 3 | 5 | 7
Not Completed | 0 | 1 | 0 | 1 | 0
Not completed — Cancel prior to treatment | 0 | 0 | 0 | 1 | 0
Not completed — Ineligible | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 0 | Dose Level 0B | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 4 | 4 | 3 | 6 | 7 | 24
Age, Continuous [Median (Full Range); unit: years] | 72.5 [59 to 81] | 62.5 [24 to 64] | 67 [47 to 67] | 63.5 [40 to 75] | 61 [58 to 69] | 63.5 [24 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 2 | 3 | 10
  Male | 3 | 1 | 2 | 4 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 4 | 3 | 6 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 0 | 2
  White | 3 | 3 | 3 | 5 | 6 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 3 | 6 | 7 | 24

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (Phase I)
Description: Dose Limiting Toxicity (DLTs) will be assessed during the first cycle of induction chemotherapy.
  The following events are considered DLTs: Grade 4 neutropenia (ANC < 500) lasting more than 14 days, Febrile neutropenia, Grade 4 thrombocytopenia, dose delay of greater than 3 weeks due to failure to recover counts, treatment-related grade 3 or grade 4 non-hematological toxicity (excluding alopecia, fatigue, hypersensitivity reaction, nausea, vomiting, constipation, diarrhea, hypokalemia, hypomagnesemia, hypocalcemia, hypophosphatemia, and grade 3 hypertension), a dose delay of greater than 3 weeks for non-hematological toxicity despite replacement of electrolytes, maximum treatment for diarrhea, nausea, vomiting, and hypertension, any drug-related death.
  The number of patients reporting a DLT are reported below. The maximum tolerated dose (MTD) will be determined as the highest dose where 1 or fewer out of 6 patients reports a DLT.
Time Frame: Up to 3 weeks
Population: Dose Level 0 was not included in this outcome due to a change in treatment regimen. On Dose Level 0B, 1 patient was ineligible based on protocol criteria. On dose level 2, 1 patient cancelled prior to treatment, 1 had a dosing error and 1 pt did not complete cycle 1. On Dose Level 3, 1 patient cancelled prior to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0 | Dose Level 0B | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Relative Change in Tumor Size as Measured by RECIST (Phase II)
Description: Treatment arms will be compared using the nonparametric Wilcoxon rank-sum test.
Time Frame: From baseline to 6 weeks
Population: The Phase II portion of this study never opened and no analysis was planned.
Groups:
- Arm II (Placebo, Combination Chemotherapy): Patients receive placebo PO BID on days 1-7. Patients also receive paclitaxel and carboplatin as in Phase I. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Within 10 days from completion of course 2, patients begin concomitant chemoradiotherapy.
  Carboplatin: Given IV
  Cisplatin: Given IV
  Fluorouracil: Given IV
  Hydroxyurea: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Placebo: Given PO
  Radiation Therapy: Undergo radiation therapy
Arm/Group | Arm I (Veliparib, Combination Chemotherapy) | Arm II (Placebo, Combination Chemotherapy)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Toxicity (Phase I and Phase II)
Description: Adverse Events were collected each cycle during treatment and follow-up according to the CTCAE v4.0 guidelines. The worst graded adverse event was determined for each patient. Below is a table of the number of patients that reported a Grade 3 or Grade 4 or Grade 5 as their worst reported event.
Time Frame: upt to 5 years
Population: All patients that started protocol treatment and were evaluated for adverse events are included in this analysis. The Phase II portion of the study never opened, and therefore no data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0 | Dose Level 0B | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 4 | 3 | 3 | 5 | 7
Participants
  Grade 3 Adverse Event | 0 | 2 | 2 | 4 | 6
  Grade 4 Adverse Event | 3 | 1 | 1 | 0 | 1
  Grade 5 Adverse Event | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: PFS (Phase II)
Description: Summarized using the method of Kaplan-Meier, and compared between groups using the log-rank test. Multivariate Cox proportional hazards regression models will be used to further explore group differences adjusting for other prognostic factors, as well as to estimate hazard ratios.
Time Frame: Up to 5 years
Population: No patients were eligible for this Phase II endpoint. The Phase II portion of this study never opened.
Arm/Group | Arm I (Veliparib, Combination Chemotherapy) | Arm II (Placebo, Combination Chemotherapy)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Disease-free Survival (Phase II)
Description: as for outcome 4
Time Frame: Up to 5 years
Population: No patients were eligible for this Phase II endpoint. The Phase II portion of this study never opened.
Arm/Group | Arm I (Veliparib, Combination Chemotherapy) | Arm II (Placebo, Combination Chemotherapy)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Local or Distant Progression (Phase II)
Description: as for outcome 4
Time Frame: Up to 5 years
Population: No patients were eligible for this Phase II endpoint. The Phase II portion of this study never opened.
Arm/Group | Arm I (Veliparib, Combination Chemotherapy) | Arm II (Placebo, Combination Chemotherapy)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: DSS (Phase II)
Description: Summarized using cumulative incidence, and will be compared between groups using Gray's test. Multivariate Cox proportional hazards regression models will be used to further explore group differences adjusting for other prognostic factors, as well as to estimate hazard ratios.
Time Frame: Up to 5 years
Population: No patients were eligible for this Phase II endpoint. The Phase II portion of this study never opened.
Arm/Group | Arm I (Veliparib, Combination Chemotherapy) | Arm II (Placebo, Combination Chemotherapy)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: OS (Phase II)
Description: as for outcome 4
Time Frame: Up to 5 years
Population: No patients were eligible for this Phase II endpoint. The Phase II portion of this study never opened.
Arm/Group | Arm I (Veliparib, Combination Chemotherapy) | Arm II (Placebo, Combination Chemotherapy)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected every week during treatment (up to 13 weeks) and then every 6 months during clinical follow-up for a maximum of 5 years from registration.
Description: Adverse events were collected every week during treatment (up to 13 weeks) and then every 6 months during clinical follow-up for a maximum of 5 years from registration. All patients that began study treatment and were assessed for adverse events are included in this analysis. Patients that cancelled or were not evaluated for adverse events were not included.
Arm/Group | Dose Level 0 | Dose Level 0B | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/3 | 0/3 | 1/3 | 0/5 | 5/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 5/5 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 (N=3) | Dose Level 0B (N=3) | Dose Level 1 (N=3) | Dose Level 2 (N=5) | Dose Level 3 (N=7)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 (N=3) | Dose Level 0B (N=3) | Dose Level 1 (N=3) | Dose Level 2 (N=5) | Dose Level 3 (N=7)
Anemia (Blood and lymphatic system disorders) | 3 (18) | 2 (7) | 3 (10) | 4 (10) | 7 (30)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hyperthyroidism (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (5) | 1 (3) | 1 (1) | 1 (2) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 3 (10) | 1 (1) | 1 (2) | 2 (3) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 1 (3) | 1 (6) | 3 (9) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 3 (14) | 1 (7) | 0 (0) | 2 (5) | 4 (12)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (24) | 3 (12) | 3 (22) | 5 (23) | 4 (24)
Nausea (Gastrointestinal disorders) | 2 (7) | 2 (8) | 3 (10) | 2 (3) | 5 (9)
Oral hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (7) | 1 (5) | 3 (10) | 3 (12) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (2) | 2 (3) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (19) | 3 (13) | 3 (16) | 3 (10) | 7 (29)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 2 (13)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (10)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 (15) | 2 (6) | 3 (14) | 3 (9) | 4 (10)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (4) | 1 (1) | 2 (2) | 5 (21) | 3 (3)
Alkaline phosphatase increased (Investigations) | 3 (8) | 1 (1) | 2 (2) | 2 (16) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 1 (1) | 2 (4) | 5 (20) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 1 (4)
Creatinine increased (Investigations) | 1 (7) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (17) | 1 (6) | 0 (0) | 2 (5) | 6 (23)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (5) | 3 (6) | 2 (5) | 4 (8) | 6 (18)
Platelet count decreased (Investigations) | 3 (10) | 3 (11) | 3 (14) | 4 (28) | 7 (16)
Serum amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 2 (3) | 0 (0) | 1 (1) | 2 (4) | 2 (6)
White blood cell decreased (Investigations) | 2 (4) | 1 (3) | 0 (0) | 3 (3) | 6 (21)
Anorexia (Metabolism and nutrition disorders) | 2 (6) | 2 (11) | 3 (5) | 3 (12) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (13) | 0 (0) | 0 (0) | 1 (1) | 5 (17)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (9) | 1 (1) | 0 (0) | 0 (0) | 1 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 1 (1) | 0 (0) | 3 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (11)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5) | 1 (4) | 0 (0) | 1 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 1 (1) | 1 (1) | 0 (0) | 3 (6)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Dysgeusia (Nervous system disorders) | 1 (2) | 3 (10) | 1 (1) | 1 (1) | 2 (6)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (12) | 2 (10) | 4 (15)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 2 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (3) | 2 (3) | 0 (0) | 4 (7)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 2 (4) | 1 (2) | 2 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT01711541/Prot_SAP_000.pdf